CLINICAL TRIAL: NCT04052139
Title: Pilot Study of Opioid-receptor Antagonists to Reduce Pain and Inflammation Among HIV-Infected Persons With Alcohol Problems
Brief Title: St. PETERsburg Pain and Alcohol Intervention With Naltrexone and Gabapentin
Acronym: UH3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-39162; UH3AA026193 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Chronic Pain; Alcohol Use, Unspecified; HIV Infections
Keywords: Pain; Alcohol; HIV; Inflammation; Low-dose naltrexone; Gabapentin
MeSH Terms: conditions — Chronic Pain; Alcohol Drinking; HIV Infections; Pain; Inflammation | interventions — Naltrexone; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose naltrexone (Active Comparator): Participants randomized to this group will receive low dose naltrexone (4.5 mg) for 8 weeks.
  Interventions: Drug: Low-dose naltrexone
- Gabapentin (Active Comparator): Participants randomized to the gabapentin arm begin on a dose of 300 mg daily (300 mg qd). In week 2, participants will take 300 mg of gabapentin three times daily. In week 3 the dose will be titrated up to 1800 mg daily (300 mg+300 mg tid) will remain on the dose until week 8, when they will be tapered back down to 900 mg daily (300 mg tid). In week 8, in days 1-4 participants will take 1800 mg daily (300 mg+300 mg tid); in days 5-7, participants will take 900 mg daily (300 mg of gabapentin three times daily).
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Participants will receive a placebo to be taken three times daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose naltrexone — 4.5 mg of low dose naltrexone taken once daily for 8 weeks. In week 1, participants will take 4.5mg of naltrexone once daily. In week 2, participants will take 4.5mg of naltrexone once daily, and a placebo capsule twice daily. In weeks 3 through 7, participants will take 1 placebo capsule with 4.5 mg mg of naltrexone once daily, and 2 placebo capsules twice daily. In week 8, in days 1-4 participants will take 4.5 mg of naltrexone with a placebo capsule once daily and 2 placebo capsules twice daily; in days 5-7, participants will take 4.5 mg of naltrexone once daily, and a placebo capsule twice daily.
  Arms: Low-dose naltrexone
Drug: Gabapentin — Dose will begin at 300 mg daily (300 mg qd), in week 2 the dose will be titrated up to 900 mg daily (300 mg tid). In week 3, the dose will be titrated to 1800 mg daily ( 2 capsules of 300 mg tid) and participants will remain on that dose until week 8. In week 8, in days 1-4 participants will take 1800 mg daily (300 mg+300 mg tid); in days 5-7, participants will take 900 mg daily (300 mg of gabapentin three times daily).
  Arms: Gabapentin
Drug: Placebo — In week 1, participants will take 1 placebo capsule once daily. In week 2, participants will take 1 placebo capsule three times per day. In weeks 3 through 7, 2 placebo capsules three times per day. In week 8, in days 1-4 participants will take 2 placebo capsules three times per day; in days 5-7, participants will take 1 placebo capsule three times per day. The placebo medications will be composed of lactose and will not contain active ingredients.
  Arms: Placebo

SUMMARY:
This study is a 3-arm pilot, randomized, double-blinded, placebo-controlled study of low-dose naltrexone and gabapentin versus placebo among HIV-positive persons with heavy alcohol use and chronic pain to provide estimates of their effects on 1) pain; 2) inflammation; and 3) measures of HIV control. Participants will be followed for 12 weeks. Assessments of study outcomes will be compared at week 8 (end of treatment phase).

DETAILED DESCRIPTION:
Pain is a common co-morbidity for HIV-positive patients.Prevalence studies suggest that, on average, half of all HIV-positive persons suffer pain. Chronic pain can lead to heavy alcohol use among HIV-positive persons, which may in turn be a barrier to treatment/control of HIV and contribute to spread of HIV. Thus there is an urgent need to address pain among persons with HIV. It is timely and relevant to conduct research on gabapentin, as it has emerged as one of the most commonly prescribed non-opioid medications for pain despite the fact that gabapentin is only FDA approved for "post-herpetic neuralgia" and the literature to support its use for generalized chronic pain is limited. And yet, gabapentin has demonstrated benefits for treatment of alcohol use disorder, and therefore, like naltrexone, it could have a specific role for treating patients with chronic pain and unhealthy alcohol use. This study is a 3-arm pilot, randomized, double-blinded, placebo-controlled study of low-dose naltrexone and gabapentin vs. placebo among HIV-positive persons with heavy alcohol use and chronic pain to provide estimates of their effects on 1) pain (both self-reported and experimental/cold pressor test; 2) inflammation (i.e., levels of inflammatory cytokines IL-6, IL-1β, IL-10, and TNF-α); and 3) measures of HIV control (CD4 count and viral load).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* HIV-positive
* Chronic pain (present ≥3 mo) of moderate to severe intensity
* Heavy drinking past year (Based on NIAAA criteria: > 14 standard drinks per week/ > 4 drinks in a day for men; > 7 drinks in the past week/ > 3 drinks in a day for women)
* If female, negative pregnancy test and willing to use adequate birth control
* Provision of contact information for 2 contacts to assist with follow-up
* Stable address within 100 kilometers of St. Petersburg
* Possession of a telephone (home or cell)
* Able and willing to comply with all study protocols and procedures

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment resulting in inability to provide informed consent based on research assessor (RA) assessment
* Known active TB or current febrile illness
* Breastfeeding
* Known uncontrolled psychiatric illness (such as active psychosis)
* Current suicidal ideation
* History of hypersensitivity to naltrexone, gabapentin, or naloxone
* Current use (past week) of illicit or prescribed opiates as documented by either self-report or positive urine drug test
* Unwilling to abstain from opiates during the treatment period
* Current use of neuroleptics
* History of seizure disorder
* Known liver failure
* AST/ALT levels >5x normal
* CrCl< 60mL/min
* History of Reynaud's disease
* Planned surgeries in the next 3 months
* Enrolled in another HIV and/or substance use medication intervention study
* Taking naltrexone in the past 30 days
* Taking gabapentin in the past 30 days
* Taking pregabalin in the past 30 days
* Diagnosis of chronic obstructive pulmonary disease (COPD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Samet, MD, MA, MPH, Principal Investigator — Boston University/Boston Medical Center
Locations (1):
- First St. Petersburg Pavlov State Medical University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
All data from the study will be placed into the URBAN ARCH repository.

REFERENCES:
- [Derived] Tsui JI, Rossi SL, Cheng DM, Bendiks S, Vetrova M, Blokhina E, Winter M, Gnatienko N, Backonja M, Bryant K, Krupitsky E, Samet JH. Pilot RCT comparing low-dose naltrexone, gabapentin and placebo to reduce pain among people with HIV with alcohol problems. PLoS One. 2024 Feb 26;19(2):e0297948. doi: 10.1371/journal.pone.0297948. eCollection 2024. PMID 38408060
- See also: URBAN ARCH, a member of NIAAA CHAART (Consortiums for HIV/AIDS & Alcohol Research Translation) initiative, conducts and disseminates interdisciplinary research on how alcohol impacts people with HIV and develops interventions to reduce related outcomes. — http://www.urbanarch.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Started | 15 | 15 | 15
4-weeks | 14 | 15 | 15
8-weeks | 12 | 15 | 15
12-weeks | 12 | 15 | 15
Completed | 12 | 15 | 15
Not Completed | 3 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (6) | 41 (7) | 41 (7) | 41 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 16
  Male | 9 | 10 | 10 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 15 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 15 | 15 | 45
Region of Enrollment [Number; unit: participants]
  Russia | 15 | 15 | 15 | 45
Education - 9 grades or more [Count of Participants; unit: Participants] | 15 | 15 | 15 | 45
Marital status [Count of Participants; unit: Participants]
  Married/living with partner/long-term relationship | 5 | 11 | 6 | 22
  Never married/divorced/widowed/separated | 10 | 4 | 9 | 23
Harmful or hazardous drinking (AUDIT) [Count of Participants; unit: Participants] — Number of participants with harmful/hazardous drinking. Measured via the Alcohol Use Disorders Identification Test (AUDIT). A score of 8 or greater refers to harmful/hazardous drinking. Scores range from 0 (abstainer) to 40.
  Participants
    AUDIT score <8 | 5 | 6 | 7 | 18
    AUDIT score 8+ | 10 | 9 | 8 | 27
Number of heavy drinking days in past 30 days [Mean (Standard Deviation); unit: days] — Mean number of heavy drinking days in past 30 days. Measured via the Timeline Follow-back for past 30 days. Heavy drinking defined as > 4 drinks in a day for men; > 3 drinks in a day for women.
  days | 2 (4) | 2 (3) | 2 (4) | 2 (4)
Past month heavy drinking days (%) [Mean (Standard Deviation); unit: % days] — Mean (%) past month heavy drinking days. Measured via the Timeline Follow-back for past 30 days. Number of heavy drinking days divided by 30. Heavy drinking defined as > 4 drinks in a day for men; > 3 drinks in a day for women.
  % days | 8 (14.6) | 6.7 (9.4) | 8 (14.5) | 7.6 (12.8)
Lifetime opioid use [Count of Participants; unit: Participants] — Number of participants who have used at least one listed opioid in their lifetime (heroin, methadone, other opioid [codeine, china white, fentanyl, Khanka] by itself, krokodil, heroin mixed with stimulants [Jeff, ephedrine, amphetamine, methamphetamine, cocaine or crack]).
  Participants
    No use of opioids in lifetime | 6 | 6 | 8 | 20
    Use of opioids in lifetime | 9 | 9 | 7 | 25
Past week pain severity [Mean (Standard Deviation); unit: units on a scale] — Mean past week pain severity (score 0 [no pain] -10 [high pain]). Pain severity will be measured using the Brief Pain Inventory
  units on a scale | 3.2 (1.4) | 3.1 (1.3) | 3.3 (1.5) | 3.2 (1.3)
Past week pain interference [Mean (Standard Deviation); unit: units on a scale] — Mean past week pain interference (score 0 [no pain] -10 [high pain]). Pain interference will be measured using the Brief Pain Inventory
  units on a scale | 3 (2) | 3 (2) | 3 (2) | 3 (2)
Cold pain threshold [Mean (Standard Deviation); unit: seconds] — Mean number of seconds until a participant feels pain while their hand in submerged in a container of iced water. Participants were instructed to let the research assessor know when they first felt pain.
  seconds | 21 (17) | 15 (13) | 14 (6) | 17 (13)
Cold pain tolerance [Mean (Standard Deviation); unit: seconds] — Mean number of seconds a participant can keep their hand submerged in a container of iced water. Participants were instructed to keep their hand in as long as they could, up to 3 minutes.
  seconds | 42 (33) | 33 (25) | 36 (41) | 37 (33)
IL-6 biomarker [Mean (Standard Deviation); unit: pg/ml] — Mean IL-6 values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
  pg/ml | 3.77 (0.66) | 3.73 (0.4) | 3.5 (0.38) | 3.67 (0.5)
IL-10 biomarker [Mean (Standard Deviation); unit: pg/ml] — Mean IL-10 values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
  pg/ml | 3.81 (0.7) | 3.85 (0.7) | 3.92 (0.8) | 3.86 (0.7)
TNF-alpha biomarker [Mean (Standard Deviation); unit: pg/ml] — Mean TNF-alpha values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
  pg/ml | 5.70 (0.7) | 5.86 (0.9) | 6.35 (1.2) | 5.97 (1.0)
IL-1-beta biomarker [Mean (Standard Deviation); unit: pg/ml] — Mean IL-1beta values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
  pg/ml | 5.73 (0.5) | 5.57 (0.7) | 5.53 (0.6) | 5.61 (0.6)
HIV viral load suppression [Count of Participants; unit: Participants] — Number of participants with suppressed HIV viral load (<250 copies/ml) and unsuppressed HIV viral load (250+ copies/ml)
  Participants
    Unsuppressed viral load | 3 | 1 | 0 | 4
    Suppressed viral load | 12 | 14 | 15 | 41
CD4 count [Mean (Standard Deviation); unit: cell/mm^3] — Mean CD4 values
  cell/mm^3 | 648 (273) | 808 (290) | 917 (381) | 791 (331)
Depressive symptoms [Count of Participants; unit: Participants] — Number of participants with depressive symptoms, measured with the Center for Epidemiologic Studies Depression Scale (CES-D). Depressive symptoms indicated as a score of 16 or above.
  Participants
    No depressive symptoms | 12 | 12 | 12 | 36
    Depressive symptoms | 3 | 3 | 3 | 9
Anxiety [Count of Participants; unit: Participants] — Number of participants with anxiety, measured with the General Anxiety Disorder-7 (GAD-7). Minimal anxiety indicated as a score of 0 to 4; mild anxiety as 5 to 9; moderate anxiety at 10 to 14; and severe anxiety at 15 to 21. Possible scores range from 0 (no anxiety) to 21.
  Participants
    Minimal anxiety | 11 | 11 | 11 | 33
    Mild anxiety | 2 | 2 | 3 | 7
    Moderate anxiety | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Past Week Pain Severity
Description: Change in past week pain severity (score 0 [no pain] -10 [high pain]) from baseline to week 8. Pain severity will be measured using the Brief Pain Inventory, which allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
units on a scale | -0.97 (0.63) | -2.12 (0.38) | -1.85 (0.61)

2. Primary Outcome: Change in Past Week Pain Interference
Description: Change in past week pain interference (score 0 [no pain]-10 [high pain]) from baseline to week 8. Pain interference will be measured using the Brief Pain Inventory, which allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
units on a scale | -1.73 (0.47) | -1.97 (0.64) | -2.14 (0.58)

3. Secondary Outcome: Change in Cold Pain Tolerance
Description: Mean change in the number of seconds a participant can keep their hand submerged in a container of iced water. Participants were instructed to keep their hand in as long as they could, up to 3 minutes.
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
seconds | -14.78 (7.61) | -3.33 (4.56) | -3.15 (6.89)

4. Secondary Outcome: Change in Percentage of Past Month Heavy Drinking Days
Description: Mean percentage of change in self-reported heavy drinking in the past 30 days of alcohol consumption obtained via the Timeline Followback (TLFB) method. The NIAAA definition of heavy drinking is used (> 4 drinks in a day for men; > 3 drinks in a day for women). Participants were asked about their alcohol consumption on each day in the previous 30 days.
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: % of change in heavy drinking days
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
% of change in heavy drinking days | 3.07 (5.17) | -4.22 (2.07) | -4.63 (4.64)

5. Secondary Outcome: Change in CD4 Count
Description: Defined as mean change in CD4 values from lab assay
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: cell/mm^3
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
cell/mm^3 | 15.85 (74.96) | -106.47 (64.94) | -52.13 (82.43)

6. Secondary Outcome: Number of Participants With a Change in HIV Viral Load Suppression Status
Description: Defined as number of participants who change from suppressed to unsuppressed or unsuppressed to suppressed from lab tests
Time Frame: Baseline, 8-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
Participants | 1 | 0 | 0

7. Secondary Outcome: Change in Biomarker IL-6
Description: Mean change in IL-6 values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
pg/ml | -0.12 (0.19) | 0.04 (0.12) | 0.29 (0.14)

8. Secondary Outcome: Change in Biomarker IL-10
Description: Mean change in IL-10 values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
pg/ml | -0.13 (0.25) | 0.07 (0.16) | -0.26 (0.23)

9. Secondary Outcome: Change in TNF-alpha
Description: Mean change in TNF-alpha values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
pg/ml | 0.27 (0.31) | 0.47 (0.15) | 0.21 (0.42)

10. Secondary Outcome: Change in IL-1beta
Description: Mean change in IL-1beta values measured on blood samples collected using commercially available enzyme-linked immunosorbent assay kits (R&D Systems).
Time Frame: Baseline, 8-weeks
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
Number analyzed (Participants) | 12 | 15 | 15
pg/ml | 0.30 (0.22) | 0.95 (0.29) | 0.41 (0.20)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline to 12 weeks.
Arm/Group | Low-dose Naltrexone | Gabapentin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 1/15
Other Adverse Events (participants affected / at risk) | 4/15 | 5/15 | 2/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Naltrexone (N=15) | Gabapentin (N=15) | Placebo (N=15)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Surgery for Acute purulent non-lactation mastitis on the left side (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose Naltrexone (N=15) | Gabapentin (N=15) | Placebo (N=15)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech impediment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sleepiness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Burning in the legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Redness of the skin of the upper body (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT04052139/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT04052139/ICF_000.pdf